CLINICAL TRIAL: NCT07102550
Title: Biliary Anastomosis in Living Donor Liver Transplant With Amniotic Tissue: A Prospective Non-Randomized Clinical Trial
Brief Title: Biliary Anastomosis in Living Donor Liver Transplant With Amniotic Tissue
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Choon Hyuck David Kwon (Other)
Responsible Party: Sponsor-Investigator, Choon Hyuck David Kwon, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-829
Record Dates: First submitted 2024-08-21; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Liver Transplant
Keywords: Living Donor Liver Transplant; Liver Transplant Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Living Donor Liver Transplant (LDLT) graft recipient (Other): LDLT recipient with MiMedx placental graft placement
  Interventions: Biological: MiMedx AmnioFix

INTERVENTIONS:
Biological: MiMedx AmnioFix — MiMedx Amniofix to be placed on biliary anastomosis of the recipient during living donor liver transplant.

SUMMARY:
The goal of this single armed, non-randomized, pilot study is to demonstrate that placental tissue grafts are safe in living donor liver transplant and assess their impact on biliary outcomes in adults.

DETAILED DESCRIPTION:
The goal of this single armed, non-randomized, pilot study is to demonstrate that placental tissue grafts are safe in living donor liver transplant and assess their impact on biliary outcomes in adults. MiMedx placental tissue grafts are registered with the FDA for homologous use in any location in the body as a protective barrier that supports the healing cascade, which is the use the investigators intend it for in this trial.

The main questions this study aims to answer are:

1. Can bile-duct reinforcement using MiMedx placental tissue grafting demonstrate equal-to-improved biliary complications in patients who are recipients of living donor liver transplant?
2. What are the rates of postoperative complications and outcomes of living donor liver transplant after using MiMedx placental tissue grafting?

Participants will:

1. undergo living donor liver transplant per standard procedures at Cleveland Clinic, including pre-procedure, post-procedure, and follow-up visits.
2. consent to the placement of MiMedx placental tissue graft around the biliary anastomosis during their liver transplant.
3. consent to allow the study team to perform a review of their medial records after each standard-of-care follow-up visit to assess presence of any biliary complications up to 1 year post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Adults >/= 18 years old
* Recipient of LDLT

Exclusion Criteria:

* Patients who are deemed unsafe for participation for any reason by our multi-disciplinary liver transplant selection committee.
* Patients < 18 years old
* Patients who cannot provide informed consent
* Patients receiving deceased donor liver transplants, or who are not undergoing Liver transplant (LT)
* Patients who do not wish to participate
* Children, cognitively-impaired persons, pregnant women, students and house staff under the direct supervision of the investigator are considered vulnerable populations and will, therefore, be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Biliary complications | 1 year post living donor liver transplant
  Biliary complications will be defined as any confirmed leakage of bile into the peritoneal cavity outside of the ductal system or biliary stricture.

SECONDARY OUTCOMES:
Post-operative Complication Rates | 1 year post living donor liver transplant
  Rates of postoperative complications and outcomes including: Re-operation, acute or chronic graft rejection, procedural intervention (in total and biliary in nature), delayed graft function, primary graft non-function, surgical site infection
Post-operative Hospital Length of Stay | From date of transplant until date of discharge from hospital, assessed up to 365 days
  Hospital length of stay
Post-operative ICU Length of Stay | From date of transplant until date of transfer out of ICU, assessed up to 365 days
  ICU length of stay (days)
Readmissions | 1 year post living donor liver transplant
  Number of readmissions post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Choon Hyuck D Kwon, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No